CLINICAL TRIAL: NCT04184908
Title: Clinical Study to Evaluate the Efectiveness and Tolerability of a New Gel for Xerostomia
Brief Title: Clinical Study New Gel for Xerostomia
Acronym: XEROSTOMIA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, UNIVERSIDAD DE MURCIA, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNIVERSITY
Record Dates: First submitted 2019-11-29; First posted 2019-12-04 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: XEROSTOMIA
Keywords: dry mouth
MeSH Terms: conditions — Xerostomia | interventions — Lubricants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP EXPERIMENTAL (Experimental): Gel xerostomia Apply 2-3 cm of the gel on the tongue, gums and oral mucosa, at least three times a day, if necessary it can be applied at night
  Interventions: Drug: gel xerostomia
- CONTROL GROUP (Placebo Comparator): Gel placebo Apply 2-3 cm of the gel on the tongue, gums and oral mucosa, at least three times a day, if necessary it can be applied at night
  Interventions: Other: gel placebo

INTERVENTIONS:
Drug: gel xerostomia — Apply 2-3 cm of the gel on the tongue, gums and oral mucosa, at least three times a day, if necessary it can be applied at night
  Other Names: lubricant and remineralizing agents
  Arms: GROUP EXPERIMENTAL
Other: gel placebo — Apply 2-3 cm of the gel on the tongue, gums and oral mucosa, at least three times a day, if necessary it can be applied at night
  Arms: CONTROL GROUP

SUMMARY:
At present, there is no single consensus protocol for the treatment of oral dryness, although the main objective is to improve the quality of life of patients. Current therapy for the control of xerostomia is based on the following measures:

1. General measures ; review and control of drugs,hydration and dietary advice:

   The main recommendations are found in the following scheme.
2. Saliva stimulants( Topics and sistemic )The option of using chewing stimuli by chewing gum with non-cariogenic sweeteners helps to improve symptoms. The investigators can also use gustatory stimuli, such as citric acid that is a potent stimulator of salivary secretion.

   Among the most commonly used pharmacological agents are: pilocarpine, bethanecol, civemiline
3. Saliva substitutes or artificial saliva. Saliva substitutes can provide a moisture retention layer in the oral mucosa and can be administered by liquids, spray, pills or gels. Topical treatments have few adverse effects and improve the quality of life of patients with xerostomia; In addition, they maintain oral health.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled clinical study to evaluate the efficacy and tolerability in patients with a non-commercialized gel and property of the promoter to treat xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes 2. Over 18 years. 3. Adequate cultural level and understanding of the clinical study. 4. Agree to voluntarily participate in the study and give their informed consent in writing 5. Present xerostomia of more than three months of evolution / sialometry less than 0.2ml / 5 min.

Exclusion criteria

The presence of at least one of the following criteria will be grounds for exclusion from the clinical trial:

1. Presence of health problems that may compromise adherence to the study protocol.
2. Pregnant or breastfeeding women.
3. Present hypersensitivity to any component of the product under study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
OHIP 14 | 1moth
  Quality of oral life. minimun 0 maximum 56 points. As it gets higher, quality of life decreases
Sialometry | 1moth
  Drenaje
Test Thonsom xerostomy | 1moth
  Xerostomia Inventory. the higher the outcome, quality of life decreases

CONTACTS AND LOCATIONS:
Locations (1):
- Lopez-Jornet Pia, Murcia, N/A = Not Applicable, Spain

REFERENCES:
- [Background] Assery MKA. Efficacy of Artificial Salivary Substitutes in Treatment of Xerostomia: A Systematic Review. J Pharm Bioallied Sci. 2019 Feb;11(Suppl 1):S1-S12. doi: 10.4103/jpbs.JPBS_220_18. PMID 30923424
- [Background] Gil-Montoya JA, Silvestre FJ, Barrios R, Silvestre-Rangil J. Treatment of xerostomia and hyposalivation in the elderly: A systematic review. Med Oral Patol Oral Cir Bucal. 2016 May 1;21(3):e355-66. doi: 10.4317/medoral.20969. PMID 27031061
- [Background] Lysik D, Niemirowicz-Laskowska K, Bucki R, Tokajuk G, Mystkowska J. Artificial Saliva: Challenges and Future Perspectives for the Treatment of Xerostomia. Int J Mol Sci. 2019 Jun 29;20(13):3199. doi: 10.3390/ijms20133199. PMID 31261876